CLINICAL TRIAL: NCT04579601
Title: Implementation of an ERAS Program in Patients Undergoing Thoracic Surgery at a Third-level University Hospital. An Ambispective Cohort Study
Brief Title: ERAS Program in Thoracic Surgery Analyzed the Effects on the Rates of Complications, Readmission and Length of Stay
Acronym: ERAS
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: EO071-18_FJD
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Thoracic Surgery
Keywords: Fast-track rehabilitation; ERAS; VATS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- ERAS group: We recruited 50 patients throughout 2018 and 2019, patients undergoing thoracic surgery within an ERAS program
  Interventions: Procedure: ERAS program
- Standard group: A group of 50 patients selected randomly prior the implementation of the ERAS program, in 2016.

INTERVENTIONS:
Procedure: ERAS program — We designed our centre's ERAS program through different measures during the preoperative, intraoperative and postoperative period. This program incluided received comprehensive multidisciplinary information, daily goals and expected discharge date, explained the expansión exercises, the video-assisted thoracoscopic surgery (VATS) under general anaesthesia combined with regional techniques, leaving only one chest tube at the end of the surgery, maintain normothermia, extubation after the end of the surgery, and early removal of the urinary catheter. From the time of extubation, the patients began oral tolerance and respiratory physiotherapy exercises. Also, the patients were allowed to walk around early.
  Groups: ERAS group

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide, representing 20,55% and 14% of cancer deaths in Spain and the United States, respectively. Currently, pulmonary resection is the treatment of choice for lung cancer. However, this surgery is associated with significant complications in almost 50% of the cases, possibly delaying patient recovery and consequently increasing hospitalisation costs.

Professor Henrik Kehlet described ERAS programs at the end of the last century. His ideas were that the application of specific measures based on scientific evidence during the perioperative period of the patient could decrease the stress produced by surgical aggression. Thus, in recent years, ERAS programs have proven effective in reducing surgical complications, length of stay and hospital costs.

Over the last years, specific ERAS surgical approaches have been described for thoracic surgery. Nevertheless, there is still a lack of evidence to support ERAS programs for pulmonary resection surgery, particularly in terms of clinical results combined with minimally invasive procedures.

Our study aims to analyze the effects of the implementation of an ERAS program in patients undergoing pulmonary resection in a tertiary university hospital on the rates of complications and readmission and the length of stay.

DETAILED DESCRIPTION:
This study analyzes the implementation of an ERAS program in a thoracic service of a third level hospital (Hospital Fundación Jiménez Díaz, Madrid, Spain). To this end, the investigators designed an ambispective cohort study, with a prospective arm of patients undergoing thoracic surgery within an ERAS program versus a retrospective arm of patients before the implementation of the protocol. Our centre's ethics committee approved our study before the start of patient recruitment, January 2018 Ref: EO071-18_FJD. This study followed the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) reporting guideline for cohort studies.

After informed consent, the investigators included patients consecutively since the implementation, except those who refused the inclusion in the study or were under 18 years old. The investigators also asked for informed consent from the patients who were part of the retrospective cohort. For the calculation of the required sample size, the investigators assumed that the ERAS program would result in a 25% reduction in the absolute risk of suffering a surgical complication. Since the surgical complication rate for our patients in 2016 was 40%, a type-I error of 5% and a power of 80% would require 47 patients per arm.

Procedures The investigators recruited 50 patients throughout 2018 and 2019 and compared them with data from the last 50 patients in 2016, the year in which the investigators knew the surgical complication rate. The investigators followed up each patient for 30 days after surgery through hospital and primary care medical records. Demographic and comorbidity data were collected from all patients, from which the investigators calculated Charlson's comorbidity index14 for all patients.

The investigators designed our centre's ERAS program through different measures during the preoperative, intraoperative and postoperative period. During the preoperative period, the patients and their families received comprehensive multidisciplinary information about the protocol, as well as their daily goals and expected discharge date. Also, a team specialized in therapy against lung diseases taught patients pulmonary expansion exercises to be carried out until surgery was performed. Smoking cessation and nutritional screening of the patient were also part of this stage.

The patients underwent video-assisted thoracoscopic surgery (VATS), whenever possible, leaving a chest tube at the end of the surgery. All subjects received antibiotic and antithrombotic prophylaxis. Intraoperative management of patients was performed under general anaesthesia combined with regional techniques for pain control, avoiding the use of benzodiazepines and opioids. Those patients in whom thoracic epidural catheter was implemented during surgery continued its use through a patient-controlled analgesia system. Besides, a hot air system warmed the patients during surgery to maintain normothermia. Extubation was performed as soon as possible after the end of the surgery, and encouraged early removal of the urinary catheter.

From the time of extubation, the patients began oral tolerance and respiratory physiotherapy exercises. Also, the patients were allowed to walk around early. The patients were discharged when they were free of complications, without severe pain, urinary catheter or chest tube.

Outcomes The primary outcome was the number of patients with 30-day surgical complications. The investigators defined air leakage, bleeding, infection, and reintervention as surgical complications. Secondary outcome included ERAS adherence, no-surgical complications, mortality, readmission, reintervention rates, pain (defined as any level of pain that prevents early ambulation) and hospital lenght of stay. To evaluate ERAS adherence, the investigators defined seven items: VATS approach, regional analgesia, oral tolerance within 6 hours, urinary catheter removal within 24 hours, ambulation within 24 hours, respiratory physiotherapy within 24 hours and chest tube removal within 48 hours.

Statistical analysis The investigators analyzed outcomes depending on whether the patient belonged to the ERAS program or the retrospective standard cohort. The discrete and continuous variables were described as number and percentage and median (interquartile range [IQR]) and their differences analyzed using the Pearson test or the Wilcoxon rank-sum tests. Subsequently, according to the adherence rate to ERAS items (regardless of whether the patients belonged to the ERAS or the retrospective standard cohort).

The investigators performed a multivariate logistic analysis to study the association of complication rates, readmission or pain with ERAS adherence, clinical and demographic data, presenting the results in forest plots as odds ratio with 95% confidence interval. Similarly, the investigators used Cox regression for multivariate analysis of length of stay, presenting the results in forest plot as hazard ratio with 95% confidence interval. To avoid errors by multiple comparisons, the investigators calculated the respective q-value for each p-value to maintain a false discovery rate below 5%.

The investigators considered comparisons in which p-value and q-value were below .05 as being statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing of a thoracic surgery during the recruitmet period with

  ->18 years
* always after informed consent.

Exclusion Criteria:

* PAtients without consent
* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After informed consent, we included patients consecutively since the implementation, except those who refused the inclusion in the study or were under 18 years old. We also asked for informed consent from the patients who were part of the retrospective cohort
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Surgical complication | 30 days
  We defined air leakage, bleeding, infection, and reintervention as surgical complications.

SECONDARY OUTCOMES:
Rate of Non surgical complication | 30 days
  Any circunstance wich increases the time of admission and is not included in the surgical complication

OTHER OUTCOMES:
ERAS Adherence | 30 days
  compliance for each of the protocol items
Mortality | 30 days
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Bellas, Principal Investigator — Institut Fundación Jiménez Díaz; Luis E Muñoz, Study Director — Instituto Fundación Jiménez Díaz
Locations (1):
- Fundación Jiménez Díaz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Demographic and comorbidity data were collected from all patients, from which we calculated Charlson's comorbidity index. Our plan is to share all the data that lead us to our results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Upon request the database will be shared, if it were to be included in another study, they would have to include us as collaborators of the same

REFERENCES:
- [Background] Das-Neves-Pereira JC, Bagan P, Coimbra-Israel AP, Grimaillof-Junior A, Cesar-Lopez G, Milanez-de-Campos JR, Riquet M, Biscegli-Jatene F. Fast-track rehabilitation for lung cancer lobectomy: a five-year experience. Eur J Cardiothorac Surg. 2009 Aug;36(2):383-91; discussion 391-2. doi: 10.1016/j.ejcts.2009.02.020. Epub 2009 Mar 26. PMID 19324571
- [Background] ERAS Compliance Group. The Impact of Enhanced Recovery Protocol Compliance on Elective Colorectal Cancer Resection: Results From an International Registry. Ann Surg. 2015 Jun;261(6):1153-9. doi: 10.1097/SLA.0000000000001029. PMID 25671587
- [Background] Muehling BM, Halter GL, Schelzig H, Meierhenrich R, Steffen P, Sunder-Plassmann L, Orend KH. Reduction of postoperative pulmonary complications after lung surgery using a fast track clinical pathway. Eur J Cardiothorac Surg. 2008 Jul;34(1):174-80. doi: 10.1016/j.ejcts.2008.04.009. Epub 2008 May 19. PMID 18490173
- [Background] Ripolles-Melchor J, Ramirez-Rodriguez JM, Casans-Frances R, Aldecoa C, Abad-Motos A, Logrono-Egea M, Garcia-Erce JA, Camps-Cervantes A, Ferrando-Ortola C, Suarez de la Rica A, Cuellar-Martinez A, Marmana-Mezquita S, Abad-Gurumeta A, Calvo-Vecino JM; POWER Study Investigators Group for the Spanish Perioperative Audit and Research Network (REDGERM). Association Between Use of Enhanced Recovery After Surgery Protocol and Postoperative Complications in Colorectal Surgery: The Postoperative Outcomes Within Enhanced Recovery After Surgery Protocol (POWER) Study. JAMA Surg. 2019 Aug 1;154(8):725-736. doi: 10.1001/jamasurg.2019.0995. PMID 31066889
- [Result] Falcoz PE, Puyraveau M, Thomas PA, Decaluwe H, Hurtgen M, Petersen RH, Hansen H, Brunelli A; ESTS Database Committee and ESTS Minimally Invasive Interest Group. Video-assisted thoracoscopic surgery versus open lobectomy for primary non-small-cell lung cancer: a propensity-matched analysis of outcome from the European Society of Thoracic Surgeon database. Eur J Cardiothorac Surg. 2016 Feb;49(2):602-9. doi: 10.1093/ejcts/ezv154. Epub 2015 Apr 26. PMID 25913824

DOCUMENTS (2):
  • Study Protocol (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT04579601/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT04579601/SAP_001.pdf